CLINICAL TRIAL: NCT02043808
Title: The Comparative Safety and Effectiveness of Warfarin and Dabigatran Utilized in the Department of Defense (DoD) Non-Valvular Atrial Fibrillation (NVAF) Patient Population-A Retrospective Database Analysis
Brief Title: The Safety and Effectiveness of Warfarin and Dabigatran Prescribed in the Non-Valvular Atrial Fibrillation Population With DoD Healthcare Coverage
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1160.183
Record Dates: First submitted 2014-01-10; First posted 2014-01-23 (Estimated); Results first posted 2015-07-03 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Dabigatran
- Warfarin

SUMMARY:
The objective is to assess the safety and effectiveness of new dabigatran and warfarin patients diagnosed with NVAF in the US DoD population.

DETAILED DESCRIPTION:
Study Design:

Retrospective

ELIGIBILITY:
Inclusion criteria:

* Patients must be continuously enrolled in a health plan during the pre-index period;
* Patients must have at least one inpatient, or one physician office visit, emergency room visit with a diagnosis of AF (ICD-9-CM diagnosis code: 427.31in any position) on the index date or during the pre-index period;
* Patients must have a prescription for dabigatran or warfarin (this first prescription will be the index date);
* Patients must be treatment naive from all OAC use prior to first dabigatran or warfarin prescription;
* Aged 18-89 on the index date;

Exclusion criteria:

* Patients with valvular procedures related to the baseline AF diagnosis will be excluded;
* Patients with transient causes of AF such as hyperthyroidism, any cardiac surgery, pericarditis, mycoarditis, pulmonary embolism within 3 months prior to their first diagnosis of AF;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NVAF
Sampling Method: Non-Probability Sample
Enrollment: 25586 (Actual)
Dates: Start 2014-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1160.183.01 Boehringer Ingelheim Investigational Site, Lexington, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Existing data cohort design with propensity score matching (PSM). Variables included in the final propensity score model were: age, gender index year, baseline CHADS(2) score, baseline CHA(2)DS(2)-VASc score, baseline HAS-BLED score, baseline use of several medications and presence of several baseline co-morbidities.
Groups:
- Dabigatran: Oral anticoagulant treatment-naive non-valvular atrial fibrillation (NVAF) patients aged 18-89 with their first prescription claim for dabigatran (either FDA-approved dose) during the study identification period (1 October 2010 and 31 July 2012).
- Warfarin: Oral anticoagulant treatment-naive non-valvular atrial fibrillation (NVAF) patients aged 18-89 with their first prescription claim for warfarin during the study identification period (1 October 2010 and 31 July 2012).
Period: Overall Study
Arm/Group | Dabigatran | Warfarin
Started | 12793 | 12793
Completed | 12793 | 12793
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Post-PSM set
Groups:
- Total: Total of all reporting groups
Arm/Group | Dabigatran | Warfarin | Total
Number analyzed (Participants) | 12793 | 12793 | 25586
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.8 (9.3) | 74.0 (9.0) | 73.9 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5277 | 5253 | 10530
  Male | 7516 | 7540 | 15056

OUTCOME MEASURES:

1. Primary Outcome: Stroke (Hemorrhagic, Ischemic)
Description: Event rate of stroke (hemorrhagic, ischemic).
  Variables in the final propensity score model: age, gender index year, baseline CHADS(2) score (Congestive heart failure, Hypertension, Age ≥75 years, Diabetes mellitus, Prior Stroke or transient ischemic attack (TIA) or Thromboembolism), baseline CHA(2)DS(2)-VASc score (Congestive heart failure, Hypertension, Age ≥75 years (doubled), Diabetes mellitus, Stroke (doubled), Vascular disease, Age 65-74 years, Sex category), baseline HAS-BLED score (Hypertension, Abnormal renal/liver function, Stroke, Bleeding history or predisposition, Labile International Normalized Ratio, Elderly, Drugs/alcohol concomitantly), baseline use of several medications and presence of several baseline co-morbidities.
  The 12-month period prior to and including the index date was defined as the baseline period. Patients were required to have an NVAF diagnosis during this baseline period.
Time Frame: From October 1, 2009 through July 31, 2013 (the study period)
Population: All patients in the post-propensity score matching cohort
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 12793 | 12793
Events per 1000 person-years | 9.15 [7.41 to 11.19] | 13.19 [10.74 to 16.05]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; Test type: Superiority or Other; Crude event rate ratio = 0.69, 95% CI 2-sided [0.52 to 0.92] — Crude event rate ratio for dabigatran with warfarin as the reference group

2. Primary Outcome: Major Bleeding
Description: Event rate of major bleeding.
  The 12-month period prior to and including the index date was defined as the baseline period. Patients were required to have an NVAF diagnosis during this baseline period.
Time Frame: From October 1, 2009 through July 31, 2013 (the study period)
Population: All patients in the post-propensity score matching cohort
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 12793 | 12793
Events per 1000 person-years | 30.84 [27.55 to 34.42] | 37.04 [32.82 to 41.65]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; Test type: Superiority or Other; Crude event rate ratio = 0.83, 95% CI 2-sided [0.71 to 0.98] — Crude event rate ratio for dabigatran with warfarin as the reference group

3. Secondary Outcome: Ischemic Stroke
Description: Event rate of ischemic stroke.
  The 12-month period prior to and including the index date was defined as the baseline period. Patients were required to have an NVAF diagnosis during this baseline period.
Time Frame: From October 1, 2009 through July 31, 2013 (the study period)
Population: All patients in the post-propensity score matching cohort
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 12793 | 12793
Events per 1000 person-years | 8.48 [6.80 to 10.45] | 10.69 [8.49 to 13.28]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; Test type: Superiority or Other; Crude event rate ratio = 0.79, 95% CI 2-sided [0.59 to 1.07] — Crude event rate ratio for dabigatran with warfarin as the reference group

4. Secondary Outcome: Hemorrhagic Stroke
Description: Event rate of hemorrhagic stroke.
  The 12-month period prior to and including the index date was defined as the baseline period. Patients were required to have an NVAF diagnosis during this baseline period.
Time Frame: From October 1, 2009 through July 31, 2013 (the study period).
Population: All patients in the post-propensity score matching cohort
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 12793 | 12793
Events per 1000 person-years | 0.77 [0.33 to 1.51] | 2.50 [1.50 to 3.90]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; Test type: Superiority or Other; Crude event rate ratio = 0.31, 95% CI 2-sided [0.13 to 0.70] — Crude event rate ratio for dabigatran with warfarin as the reference group

5. Secondary Outcome: Major Intracranial Bleeding
Description: Event rate of major intracranial bleeding.
  The 12-month period prior to and including the index date was defined as the baseline period. Patients were required to have an NVAF diagnosis during this baseline period.
Time Frame: From October 1, 2009 through July 31, 2013 (the study period).
Population: All patients in the post-propensity score matching cohort
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 12793 | 12793
Events per 1000 person-years | 2.69 [1.79 to 3.88] | 5.65 [4.09 to 7.62]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; Test type: Superiority or Other; Crude event rate ratio = 0.48, 95% CI 2-sided [0.30 to 0.77] — Crude event rate ratio for dabigatran with warfarin as the reference group

6. Secondary Outcome: Major Extracranial Bleeding
Description: Event rate of major extracranial bleeding.
  The 12-month period prior to and including the index date was defined as the baseline period. Patients were required to have an NVAF diagnosis during this baseline period.
Time Frame: From October 1, 2009 through July 31, 2013 (the study period).
Population: All patients in the post-propensity score matching cohort
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 12793 | 12793
Events per 1000 person-years | 28.13 [24.99 to 31.55] | 31.30 [27.44 to 35.56]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; Test type: Superiority or Other; Crude event rate ratio = 0.90, 95% CI 2-sided [0.76 to 1.07] — Crude event rate ratio for dabigatran with warfarin as the reference group

7. Secondary Outcome: Major GI Bleeding
Description: Event rate of major gastrointestinal (GI) bleeding.
  The 12-month period prior to and including the index date was defined as the baseline period. Patients were required to have an NVAF diagnosis during this baseline period.
Time Frame: From October 1, 2009 through July 31, 2013 (the study period).
Population: All patients in the post-propensity score matching cohort
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 12793 | 12793
Events per 1000 person-years | 25.40 [22.42 to 28.66] | 23.69 [20.34 to 27.42]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; Test type: Superiority or Other; Crude event rate ratio = 1.07, 95% CI 2-sided [0.89 to 1.30] — Crude event rate ratio for dabigatran with warfarin as the reference group

8. Secondary Outcome: Major Upper GI Bleeding
Description: Event rate of major upper gastrointestinal (GI) bleeding.
  The 12-month period prior to and including the index date was defined as the baseline period. Patients were required to have an NVAF diagnosis during this baseline period.
Time Frame: From October 1, 2009 through July 31, 2013 (the study period).
Population: All patients in the post-propensity score matching cohort
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 12793 | 12793
Events per 1000 person-years | 5.48 [4.15 to 7.10] | 7.63 [5.80 to 9.87]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; Test type: Superiority or Other; Crude event rate ratio = 0.72, 95% CI 2-sided [0.50 to 1.03] — Crude event rate ratio for dabigatran with warfarin as the reference group

9. Secondary Outcome: Major Lower GI Bleeding
Description: Event rate of major lower gastrointestinal (GI) bleeding.
  The 12-month period prior to and including the index date was defined as the baseline period. Patients were required to have an NVAF diagnosis during this baseline period.
Time Frame: From October 1, 2009 through July 31, 2013 (the study period).
Population: All patients in the post-propensity score matching cohort
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 12793 | 12793
Events per 1000 person-years | 20.25 [17.60 to 23.18] | 16.38 [13.62 to 19.52]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; Test type: Superiority or Other; Crude event rate ratio = 1.24, 95% CI 2-sided [0.99 to 1.54] — Crude event rate ratio for dabigatran with warfarin as the reference group

10. Secondary Outcome: Major Urogenital Bleeding
Description: Event rate of major urogenital bleeding.
  The 12-month period prior to and including the index date was defined as the baseline period. Patients were required to have an NVAF diagnosis during this baseline period.
Time Frame: From October 1, 2009 through July 31, 2013 (the study period).
Population: All patients in the post-propensity score matching cohort
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 12793 | 12793
Events per 1000 person-years | 1.06 [0.53 to 1.89] | 3.02 [1.92 to 4.54]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; Test type: Superiority or Other; Crude event rate ratio = 0.35, 95% CI 2-sided [0.17 to 0.72] — Crude event rate ratio for dabigatran with warfarin as the reference group

11. Secondary Outcome: Major Other Bleeding
Description: Event rate of major other bleeding.
  The 12-month period prior to and including the index date was defined as the baseline period. Patients were required to have an NVAF diagnosis during this baseline period.
Time Frame: From October 1, 2009 through July 31, 2013 (the study period).
Population: All patients in the post-propensity score matching cohort
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 12793 | 12793
Events per 1000 person-years | 1.92 [1.17 to 2.97] | 5.13 [3.65 to 7.01]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; Test type: Superiority or Other; Crude event rate ratio = 0.37, 95% CI 2-sided [0.22 to 0.64] — Crude event rate ratio for dabigatran with warfarin as the reference group

12. Secondary Outcome: Transient Ischemic Attack
Description: Event rate of transient ischemic attacks.
  The 12-month period prior to and including the index date was defined as the baseline period. Patients were required to have an NVAF diagnosis during this baseline period.
Time Frame: From October 1, 2009 through July 31, 2013 (the study period).
Population: All patients in the post-propensity score matching cohort
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 12793 | 12793
Events per 1000 person-years | 4.62 [3.40 to 6.12] | 5.53 [3.99 to 7.48]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; Test type: Superiority or Other; Crude event rate ratio = 0.83, 95% CI 2-sided [0.55 to 1.26] — Crude event rate ratio for dabigatran with warfarin as the reference group

13. Secondary Outcome: Myocardial Infarction
Description: Event rate of myocardial infarction.
  The 12-month period prior to and including the index date was defined as the baseline period. Patients were required to have an NVAF diagnosis during this baseline period.
Time Frame: From October 1, 2009 through July 31, 2013 (the study period).
Population: All patients in the post-propensity score matching cohort
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 12793 | 12793
Events per 1000 person-years | 5.09 [3.82 to 6.66] | 7.77 [5.92 to 10.03]
Statistical Analysis 1: Comparison: Dabigatran; Test type: Superiority or Other; Crude event rate ratio = 0.66, 95% CI 2-sided [0.45 to 0.95] — Crude event rate ratio for dabigatran with warfarin as the reference group

14. Secondary Outcome: Venous Thromboembolism
Description: Event rate of venous thromboembolism.
  The 12-month period prior to and including the index date was defined as the baseline period. Patients were required to have an NVAF diagnosis during this baseline period.
Time Frame: From October 1, 2009 through July 31, 2013 (the study period).
Population: All patients in the post-propensity score matching cohort
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 12793 | 12793
Events per 1000 person-years | 1.34 [0.73 to 2.25] | 2.10 [1.20 to 3.42]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; Test type: Superiority or Other; Crude event rate ratio = 0.64, 95% CI 2-sided [0.31 to 1.31] — Crude event rate ratio for dabigatran with warfarin as the reference group

15. Secondary Outcome: Deep Vein Thrombosis
Description: Event rate of deep vein thrombosis.
  The 12-month period prior to and including the index date was defined as the baseline period. Patients were required to have an NVAF diagnosis during this baseline period.
Time Frame: From October 1, 2009 through July 31, 2013 (the study period).
Population: All patients in the post-propensity score matching cohort
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 12793 | 12793
Events per 1000 person-years | 0.58 [0.21 to 1.25] | 1.31 [0.63 to 2.42]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; Test type: Superiority or Other; Crude event rate ratio = 0.44, 95% CI 2-sided [0.16 to 1.21] — Crude event rate ratio for dabigatran with warfarin as the reference group

16. Secondary Outcome: Pulmonary Embolism
Description: Event rate of pulmonary embolism.
  The 12-month period prior to and including the index date was defined as the baseline period. Patients were required to have an NVAF diagnosis during this baseline period.
Time Frame: From October 1, 2009 through July 31, 2013 (the study period).
Population: All patients in the post-propensity score matching cohort
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 12793 | 12793
Events per 1000 person-years | 0.77 [0.33 to 1.51] | 0.79 [0.29 to 1.72]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; Test type: Superiority or Other; Crude event rate ratio = 0.97, 95% CI 2-sided [0.34 to 2.81] — Crude event rate ratio for dabigatran with warfarin as the reference group

17. Secondary Outcome: Death
Description: Event rate of death, due to any cause.
  The 12-month period prior to and including the index date was defined as the baseline period. Patients were required to have an NVAF diagnosis during this baseline period.
Time Frame: From October 1, 2009 through July 31, 2013 (the study period).
Population: All patients in the post-propensity score matching cohort
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 12793 | 12793
Events per 1000 person-years | 31.28 [27.98 to 34.87] | 52.41 [47.40 to 57.82]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; Test type: Superiority or Other; Crude event rate ratio = 0.60, 95% CI 2-sided [0.52 to 0.69] — Crude event rate ratio for dabigatran with warfarin as the reference group

ADVERSE EVENTS:
Description: This is a retrospective observational study, therefore all patient data was de-identified and analysed in aggregate. Thus, individual patient data is not available and reporting of adverse events is not applicable.
Arm/Group | Dabigatran | Warfarin
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.